CLINICAL TRIAL: NCT00481611
Title: A Cross-Sectional Study of Occupational Exposure to Trichloroethylene, Chromosomal Aberrations, and Related Biomarkers in Guangdong, China
Brief Title: Cancer Markers Associated With Occupational Exposure to Trichloroethylene
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906176; 06-C-N176; NCT00353132 (obsolete NCT alias); NCT01338194 (obsolete NCT alias)
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Industrial Hygiene; Epidemiology; Neoplasms
Keywords: Industry Hygiene; Molecular Epidemiology; Cancer Susceptibility; Genotoxicity; Immune Function; Cancer Susceptability
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Red blood cells, whole blood, cryopreserved lymphocytes, cryopreserved granulocytes, FISH cells, FISH slides, RNAlater, supernatant, buccal pellets, buccal slides, serum, clot, LeukLock, buffy coat, urine.

SUMMARY:
Background:

* Trichloroethylene (TCE) is a solvent used in many medical and industrial processes.
* TCE is a carcinogen (causes cancer) in rats, but its carcinogenicity in humans is unclear. There is some evidence of increased liver and kidney cancers and of an association with non-Hodgkin lymphoma in studies of workers exposed to TCE.
* The carcinogenicity and regulation of TCE is a matter of continuing debate.

Objectives:

* To determine if TCE exposure is associated with higher levels of genetic aberrations in certain white blood cells called lymphocytes.
* To determine if TCE exposure affects lymphocyte subsets and levels of certain hormones called cytokines.

Eligibility: Workers exposed to two different levels of exposure to TCE and unexposed workers in Guangdong Province, China.

Design:

* 45 workers exposed to more than 25 parts per million (ppm) TCE, 30 workers exposed to from 10 to less than 25 ppm TCE and 45 unexposed workers will be enrolled.
* Subjects wear small instruments at work that measure chemicals in the air for 1 or 2 days during the 2-week study period. Exposed workers also wear several small skin patches on one of the two days.
* Subjects provide blood and urine samples.
* Subjects answer a questionnaire about work, smoking and drinking, use of medicines, medical history, general health, hobbies, and exposure to radiation and exposure to various substances at home.

DETAILED DESCRIPTION:
Trichloroethylene (TCE) is an industrial solvent used in degreasing, dry cleaning, and numerous other medical and industrial processes. It is a ubiquitous environmental contaminant of drinking water and is present in many EPA Superfund sites. TCE is a rodent carcinogen but its carcinogenicity in humans is unclear. There is some evidence for an elevation in liver and kidney cancers and somewhat more convincing evidence of an association with non-Hodgkin lymphoma (NHL) in epidemiological studies of occupationally exposed cohorts. Overall, the carcinogenicity of TCE and its regulation is a matter of continuing debate despite an extensive database of in vitro and in vivo animal studies and several cohort and case-control studies. IARC categorizes TCE as a probable human carcinogen. In order to address questions about TCE's potential carcinogenicity and mechanism of action in humans, we propose to conduct a cross-sectional study of early biologic effect biomarkers of genotoxicity and immunotoxicity in 45 workers exposed to greater than 25 ppm TCE, 30 workers exposed to 10-25 ppm TCE, and 45 unexposed controls in Guangdong Province, China. We will assess TCE exposure level quantitatively, collect other exposure information through a questionnaire, collect biological samples, and assay a series of biomarkers of susceptibility, intermediate and early biologic effects. Our primary goal is to determine if TCE exposure increases chromosomal aberrations in peripheral lymphocytes, with a secondary goal of determining if TCE alters levels of key cytokines in plasma and changes lymphocyte subset ratios. In addition, our collaborators at UC Berkeley will apply a new generation of cytogenetic and molecular techniques to study TCE's ability to cause specific types of chromosomal aberrations that have been associated with NHL and related hematological malignancies as well as the impact of TCE on mRNA expression and the proteome. The work will compliment previous and ongoing OEEB studies of populations exposed to TCE and has the potential to make an important contribution to what little is known about the early biologic effects of TCE in humans.

ELIGIBILITY:
* INCLUSION CRITERIA:

A total of 45 workers exposed to greater than 25 ppm TCE, 30 workers exposed from 10 to less than 25 ppm TCE, and 45 unexposed workers will be enrolled.

We will identify 45 workers from 3 factories who are exposed to greater than 25 ppm TCE. Our colleagues at the Guangdong NPCC will visit potential study factories and carry out air measurements for TCE, epichlorhydrin, methylene chloride, perchloroethylene and benzene. Factories will be selected that use only TCE for degreasing processes, have minimal co-exposures present in the same part of the workplace where TCE is used, and have used a stable manufacturing process for the past five years.

Workers will be chosen who work in part of the factory with TCE exposure, have worked for at least one year in the factory doing the same job in the same part of the manufacturing process, and have not been exposed to other genotoxic, hematotoxic, or immunotoxic compounds in any workplace. We will enroll 45 controls, who have no history of occupational exposure to TCE or to any other genotoxic, hematotoxic or immunotoxic chemicals.

EXCLUSION CRITERIA:

History of cancer, chemotherapy with DNA-damaging or immunotoxic agents, and medical treatment with ionizing radiation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We carried out a cross-sectional study of workers currently exposed to TCE in the six study factories with TCE cleaning operations and unexposed controls. Control workers were enrolled from two clothes manufacturing factories, one food production factory and a hospital that did not use TCE and were in the same geographic region as the factories that used TCE. Exclusion criteria for both TCE-exposed and control workers were history of cancer, chemotherapy and radiotherapy, as well as previous occupations with notable exposure to benzene, butadiene, styrene and/or ionizing radiation.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2006-06-15 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Hematotoxicity change | 2006-2034
  The primary goal of the study is to determine if TCE exposure is associated with higher levels of chromosomal aberrations in peripherallymphocytes. The additional goals of the study, to be funded by extramural collaborators, are to evaluate TCE urinary metabolite patterns, alterations in specific types of chromosomal aberrations that have been detected in NHL and other hematopoietic malignancies, and alterations in mRNA expression and the proteome.
Immune function | 2006-2034
  A secondary goal of the study is to determine if TCE exposure alters plasma cytokine levels and lymphocyte subsets.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Lan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Guangdong National Poison Control Center (NPCC), Guangzhou, China